CLINICAL TRIAL: NCT03078179
Title: Effect of Lactobacillus Rhamnosus GG and Bifidobacterium Longum in Children Aged 3 to 5 Years of Villavicencio and Pasto
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cooperative University of Colombia (Other)
Collaborators: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: ID 1532
Record Dates: First submitted 2017-03-03; First posted 2017-03-13 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-06

CONDITIONS: Caries, Dental
Keywords: Probiotic; Child; Care, dental
MeSH Terms: conditions — Dental Caries | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Commercial Cow Milk with Probiotic (Experimental): Probiotic enriched cow milk:
  200 ml of commercial nutritive milk fortified with probiotic Lactobacillus rhamnosus and Bifidobacterium longum once a day.
  Interventions: Dietary Supplement: Commercial Cow Milk with Probiotic
- Commercial Dairy Cow Milk (Placebo Comparator): 200 ml of commercial nutritive milk without probiotic, once a day,
  Interventions: Dietary Supplement: Commercial Dairy Cow Milk

INTERVENTIONS:
Dietary Supplement: Commercial Dairy Cow Milk — After obtaining parent´s informed consent and the baseline examination, from 3 to 5 years old, will start commercial dairy cow milk intake without probiotic (placebo) for 3 months. Clinical and microbiological testing of saliva at baseline and at the end will be performed. Differences in salivary pH (before and after a sugar solution), remineralization and demineralization in early Stage Decay and quantification of Streptococci of the mutans group.
  Arms: Commercial Dairy Cow Milk
Dietary Supplement: Commercial Cow Milk with Probiotic — The children will initiate the milk intake with probiotic one week after having ingested the milk without probiotics. They will drink the milk with probiotic for 3 months. Clinical and microbiological testing of saliva will be performed. Clinical and microbiological testing of saliva at baseline and at the end will be performed. Differences in salivary pH (before and after a sugar solution), remineralization and demineralization in early Stage Decay and quantification of Streptococci of the mutans group.
  Arms: Commercial Cow Milk with Probiotic

SUMMARY:
The objective of this pilot study is to determine if the presence of bacteria with probiotic characteristics (Lactobacillus rhamnosus GG and Bifidobacterium longum) in a commercial milk, control some measures that indicate cariogenic processes.

DETAILED DESCRIPTION:
Dental caries is a disease caused by a shift in pH balance, resulting in the formation of a biofilm composed mainly of cariogenic microflora. The interaction between this microflora and host factors conditions the deceleration or acceleration of the disease. Some biotechnology tools have been tried based on all this research, including probiotics, intended for a selective control of the etiological agents of caries and the maintenance of oral homeostasis.

Methodology: In this study, preschool children belonging to public preschool in Villavicencio and Pasto, Colombia will be invited to participate. After obtaining parent´s informed consent, the children will start commercial milk (nanPro3 Nestlé) intake without probiotic for 3 months. One week after, they will start commercial milk with probiotic during others 3 months. Clinical and microbiological testing of saliva at baseline, 3 m, and 6m will be performed. Differences in salivary pH (before and after a sugar solution), remineralization and demineralization in early Stage Decay and Established decay tooth (according to ICDAS) and quantification of Streptococci of the mutans group. Expected results: Statistically significant decrease in pH drop, demineralization in decay tooth and quantification of Streptococci of the mutans group.

ELIGIBILITY:
Inclusion Criteria:

* Pre-school children from age 3 to 5.
* Healthy children from a general health perspective, with early stage decay and established decay

Exclusion Criteria:

* Children with systemic disorders who need special care and / or who have intolerance to milk drinks or allergy to any of the components of the experimental and / or placebo beverage.
* Children who don't like milk.
* Children whit severe decay

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2017-08-20 (Actual); Study Completion 2018-05-05 (Actual)

PRIMARY OUTCOMES:
Change in remineralization of tooth decay | 3 months
  DIAGNOdent peak reading in three moments,at the beginning and at the end of the milk without probiotic (after 3 months), and at the end of the milk with probiotic (after 3 months)

SECONDARY OUTCOMES:
Change of pH of saliva before and after a rinse with sugar. | 3 months
  Saliva pH test in three moments,at the beginning and at the end of the milk without probiotic (after 3 months), and at the end of the milk with probiotic (after 3 months).
Change of Dental Plaque Index | 3 months
  Silness-Löe plaque index n three moments,at the beginning and at the end of the milk without probiotic (after 3 months), and at the end of the milk with probiotic (after 3 months).
Change of concentration of group mutans streptococci in saliva | 3 months
  Co(after 3 months).lony Forming Units (CFUs) determination in three moments,at the beginning and at the end of the milk without probiotic (after 3 months), and at the end of the milk with probiotic

CONTACTS AND LOCATIONS:
Overall Officials: María del Pilar Angarita, PhD, Principal Investigator — Cooperative University of Colombia
Locations (3):
- Colombia (3):
  - Hogar Infantil 20 de Julio, Villavicencio, Meta Department
  - Hogar Infantil La Esperanza, Villavicencio, Meta Department
  - Cdi Nidos Nutrir, Pasto

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ahola AJ, Yli-Knuuttila H, Suomalainen T, Poussa T, Ahlstrom A, Meurman JH, Korpela R. Short-term consumption of probiotic-containing cheese and its effect on dental caries risk factors. Arch Oral Biol. 2002 Nov;47(11):799-804. doi: 10.1016/s0003-9969(02)00112-7. PMID 12446187
- [Background] Aminabadi NA, Erfanparast L, Ebrahimi A, Oskouei SG. Effect of chlorhexidine pretreatment on the stability of salivary lactobacilli probiotic in six- to twelve-year-old children: a randomized controlled trial. Caries Res. 2011;45(2):148-54. doi: 10.1159/000325741. Epub 2011 Mar 31. PMID 21454978
- [Background] Twetman L, Larsen U, Fiehn NE, Stecksen-Blicks C, Twetman S. Coaggregation between probiotic bacteria and caries-associated strains: an in vitro study. Acta Odontol Scand. 2009;67(5):284-8. doi: 10.1080/00016350902984237. PMID 19479452
- [Result] Nase L, Hatakka K, Savilahti E, Saxelin M, Ponka A, Poussa T, Korpela R, Meurman JH. Effect of long-term consumption of a probiotic bacterium, Lactobacillus rhamnosus GG, in milk on dental caries and caries risk in children. Caries Res. 2001 Nov-Dec;35(6):412-20. doi: 10.1159/000047484. PMID 11799281

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT03078179/Prot_SAP_000.pdf